CLINICAL TRIAL: NCT03710200
Title: Breads Made With Triticum Heritage Varieties: Effect on Post-prandial Glycemia and Insulinemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Parma (Other)
Responsible Party: Principal Investigator, Francesca Scazzina Ph.D., Assistant Professor, University of Parma
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: BIO2
Record Dates: First submitted 2018-10-15; First posted 2018-10-18 (Actual); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Dietary Modification

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Bologna 00+S. cerevisiae yeast (Active Comparator): Bread made with Bologna flour (type 00) (modern variety)+S. cerevisiae yeast
  Interventions: Other: Bologna 00+S. cerevisiae yeast
- Bologna 1+S. cerevisiae yeast (Experimental): Bread made with Bologna flour (type 1) (modern variety)+S. cerevisiae yeast
  Interventions: Other: Bologna 1+S. cerevisiae yeast
- Bio2+S. cerevisiae yeast (Experimental): Bread made with mix Bio2 flour (type 1) (heritage mix varieties)+S. cerevisiae yeast
  Interventions: Other: Bio2+S. cerevisiae yeast
- ICARDA+S. cerevisiae yeast (Experimental): Bread made with Icarda mix (type 1) (heritage mix varieties)+S. cerevisiae yeast
  Interventions: Other: ICARDA+S. cerevisiae yeast
- Bologna 1+sourdough (Experimental): Bread made with Bologna flour (type 1) (modern variety)+sourdough
  Interventions: Other: Bologna 1+sourdough
- Bio2+sourdough (Experimental): Bread made with mix Bio2 flour (type 1) (heritage mix varieties)+sourdough
  Interventions: Other: Bio 2+sourdough
- ICARDA+sourdough (Experimental): Bread made with mix Icarda flour (type 1) (heritage mix varieties)+sourdough
  Interventions: Other: ICARDA+sourdough
- Grossi+sourdough (Experimental): Bread made with mix Grossi flour (type 1) (heritage mix varieties)+sourdough
  Interventions: Other: Grossi+sourdough

INTERVENTIONS:
Other: Bologna 00+S. cerevisiae yeast — Bologna 00 bread made with yeast (portion corresponding to 50g available carbohydrates) +500 mL of water
  Arms: Bologna 00+S. cerevisiae yeast
Other: Bologna 1+S. cerevisiae yeast — Bologna 1 bread made with yeast (portion corresponding to 50g available carbohydrates) +500 mL water
  Arms: Bologna 1+S. cerevisiae yeast
Other: Bio2+S. cerevisiae yeast — Bio2 bread made with yeast (portion corresponding to 50g available carbohydrates) +500 mL water
  Arms: Bio2+S. cerevisiae yeast
Other: ICARDA+S. cerevisiae yeast — Icarda bread made with yeast (portion corresponding to 50g available carbohydrates) +500 mL water
  Arms: ICARDA+S. cerevisiae yeast
Other: Bologna 1+sourdough — Bologna 1 bread made with sourdough (portion corresponding to 50g available carbohydrates) +500 mL water
  Arms: Bologna 1+sourdough
Other: Bio 2+sourdough — 109g of Bio2 bread made with sourdough (portion corresponding to 50g available carbohydrates) +500 mL water
  Arms: Bio2+sourdough
Other: ICARDA+sourdough — Icarda bread made with sourdough (portion corresponding to 50g available carbohydrates) +500 mL water
  Arms: ICARDA+sourdough
Other: Grossi+sourdough — Grossi bread made with sourdough (portion corresponding to 50g available carbohydrates) +500 mL water
  Arms: Grossi+sourdough

SUMMARY:
Wheat is one of the most important crop for humans and it represents a source of multiple nutrients, dietary fiber and bioactive compounds, especially if consumed as wholegrain. Several studies have suggested that Triticum heritage varieties could present a healthier and better nutritional profile than modern wheats, by providing more vitamins, minerals and nutraceutical compounds. Although the effect of ancient grain consumption have been partially investigated in both animal and human studies, the potential impact of Triticum heritage varieties compared to modern ones on post-prandial glucose metabolism is still unclear. Thus, the aim of the study was to evaluate the impact on post-prandial glycaemia and insulinemia of different types of breads formulated with flours derived from mix of heritage varieties belonging to the Triticum genus selected and cultivated in specific areas of Emilia Romagna region, compared to breads made with conventional/modern wheat flours.

DETAILED DESCRIPTION:
Cereal grain based products constitute a major part of the daily diet, and wheat is the most important crop for humans representing a source of multiple nutrients, dietary fiber and bioactive compounds, especially if consumed as wholegrain. Depending on its physical and chemicals properties, such as structure of grains, granular size of semolina, quantity and quality of fiber and phytochemicals, amylose/amylopectin ratio, wheat may vehicle protective effects on human health. After the Green Revolution, most of wheat species grown are hybrids, which derive from ancient wheat over the last 100 to 150 years. The main results of this revolution were the development of modern varieties characterized by higher yield, a reduced susceptibility to disease and insects, an increase tolerance to environmental stresses, a homogeneous maturation and a better gluten quality, compared to ancient wheat. At the same time, a decrease in genetic variability as well as a gradual depletion of the nutritional and nutraceutical properties of the wheat occurred. However, over the last years, the increase of diet-related chronic disease led to the nutritional improvement of wheat for ameliorating its health potential. Nowadays, the higher value of whole grains than refined grains is recognized, while the nutritional effects of ancient versus modern grains is still controversial. Generally, ancient species are higher in vitamins, such as folate, niacin and vitamin B6, as well as in minerals such as calcium, iron, magnesium and phosphor compared to modern species, however evidence linked to their real health in vivo effects is still lacking. Therefore, the aim of the present study is to evaluate the nutritional profile of eight breads made with ancient (Triticum heritage varieties) or modern grains on the plasma response of glucose and insulin.

ELIGIBILITY:
Inclusion Criteria:

-generally healthy

Exclusion Criteria:

* BMI≥30kg/m2
* have any health conditions (including anemia and metabolic conditions such as hypertension, dyslipidemia, impaired glucose intolerance or diabetes)
* have celiac disease
* currently taking any prescription medication for chronic diseases (including psychiatric) dietary supplements affecting the metabolism
* Women who are pregnant or breastfeeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-10-12 (Actual); Primary Completion 2018-11-15 (Actual); Study Completion 2018-11-15 (Actual)

PRIMARY OUTCOMES:
Post-prandial glycemic response | 2 hours (-10 and 0 -fasting-, 15, 30, 45, 60, 90, 120 minutes)
  Post-prandial glycemic response (iAUC)

SECONDARY OUTCOMES:
Post-prandial response for insulin | 2 hours (-10 and 0 -fasting-, 15, 30, 45, 60, 90, 120 minutes)
  Post-prandial response for insulin (iAUC)
Maximum peak for glucose and insulin | 2 hours (-10 and 0 -fasting-, 15, 30, 45, 60, 90, 120 minutes)
  maximum value of postprandial glucose and insulin response

OTHER OUTCOMES:
Satiety using a 100cm visual analog scale [ Time Frame: 2 hours ] | 2 hours
  differences in subject-rated satiety using a 100cm visual analog scale
Gastrointestinal Symptoms using a questionnaire [ Time Frame: 2 hours ] | 2 hours
  differences in subject-rated gastrointestinal symptom questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Food and Drugs, University of Parma, Parma, Italy

IPD SHARING:
Plan to Share IPD: No